CLINICAL TRIAL: NCT03963232
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Galcanezumab in Patients With Episodic Migraine-the Persist Study
Brief Title: A Study of Galcanezumab (LY2951742) in Participants With Episodic Migraine
Acronym: PERSIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17054; I5Q-MC-CGAX (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-05-16; First posted 2019-05-24 (Actual); Results first posted 2022-08-19 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Episodic Migraine
Keywords: prevention; prophylactic
MeSH Terms: interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): * Double-blind treatment phase: Participants received placebo once per month subcutaneously (SC) for 3 months.
  * Open-label treatment phase: After completion of double-blind phase, participants could enter open-label treatment phase where they received 240 milligram (mg) loading dose of galcanezumab SC (2 injections of 120 mg) in the first month followed by 120 mg per month for 2 months.
  * Follow-up phase: After completion or discontinuation from double-blind or open-label treatment phases, participants entered follow-up phase where they were observed for 4 months. No treatments administered.
  Interventions: Drug: Placebo
- Galcanezumab 120 mg (Experimental): * Double-blind treatment phase: Participants received 240 mg loading dose of galcanezumab SC (2 injections of 120 mg) in the first month followed by 120 mg per month for 2 months.
  * Open-label treatment phase: After completion of double-blind phase, participants could enter open-label treatment phase where they continued to receive 120 mg galcanezumab SC per month for 3 months.
  * Follow-up phase: After completion or discontinuation from double-blind or open-label treatment phases, participants entered follow-up phase where they were observed for 4 months. No treatments administered.
  Interventions: Drug: Galcanezumab

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742
  Arms: Galcanezumab 120 mg
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The reason for this study is to see if the drug galcanezumab is safe and effective in participants with episodic migraine. The study will last about 53 weeks and may include up to 12 visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of migraine as defined by International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 (1.1 or 1.2) (ICHD-3 2018) with a history of migraine of at least 1 year prior to screening and migraine onset prior to age 50
* Prior to screening, participants must have a history of 4-14 migraine headache days and at least 2 migraine attacks per month on average within the past 3 months

Exclusion Criteria:

* Are currently enrolled in any other clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Current use or prior exposure to galcanezumab or another calcitonin gene-related peptide (CGRP) antibody, including those who have previously completed or withdrawn from this study or any other study investigating a CGRP antibody
* Participants who are taking, or are expected to take, therapeutic antibodies during the course of the study (for example, adalimumab, infliximab, trastuzumab, bevacizumab, etc.)
* Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins, or to galcanezumab
* Women who are pregnant or nursing
* History of chronic migraine, daily persistent headache, cluster headache, medication overuse headache, migraine with brainstem aura, or hemiplegic migraine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- China (26):
  - Xuanwu Hospital-Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou
  - The First Affiliated Hospital of Zhengzhou Universtiy, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Tongji Hosp Tongji Med Col Huazhong Univ of Sci & Tech, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Affliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - No.2 Hospital Affiliated to Jilin University, Changchun, Jilin
  - Tianjin Huanhu Hospital, Tianjin, Jinnan District
  - Jiangsu Province Hospital, Nanjing, Nanjing
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - People's hospital of Rizhao, Rizhao, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - HuaShan Hospital Affiliated To Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Bao Tou Central Hospital, Baotou, Zizhiqu
- India (10):
  - Apollo Hospitals International Ltd., Ahmedabad, Gujarat
  - Artemis Hospital, Gurgaon, Haryana
  - Mangala Hospitals & Mangala Kidney Foundation, Mangalore, Karnataka
  - CHL - Apollo Hospital, Indore, Madh Prad
  - Getwell Hospital & Research Institute, Nagpur, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Gobind Ballabh Pant Hospital, New Delhi
- Russia (4):
  - First Moscow State Medical University n.a. Sechenov, Moscow
  - University Headache Clinic, Moscow
  - OOO "Medis", Nizhny Novgorod
  - Academician I.P. Pavlov First St-Petersburg State Medical University, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Zhou J, Zhong L, Chowdhury D, Skorobogatykh K, Luo G, Yang X, Zhang M, Sun L, Liu H, Qian C, Yu S. Galcanezumab in patients with episodic migraine: results from the open-label period of the phase 3 PERSIST study. J Headache Pain. 2023 Aug 4;24(1):103. doi: 10.1186/s10194-023-01613-1. PMID 37542222
- [Derived] Hu B, Li G, Li X, Wu S, Yu T, Li X, Zhao H, Jia Z, Zhuang J, Yu S. Galcanezumab in episodic migraine: the phase 3, randomized, double-blind, placebo-controlled PERSIST study. J Headache Pain. 2022 Jul 28;23(1):90. doi: 10.1186/s10194-022-01458-0. PMID 35896988
- See also: A Study of Galcanezumab (LY2951742) in Participants With Episodic Migraine — https://trials.lillytrialguide.com/en-US/trial/31dBGbS2DbVt4INep01n59

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to be conducted in three phases: a 3-month double-blind treatment phase, an optional 3-month open-label treatment phase and a 4-month follow-up phase.
Groups:
- Placebo: * Double-blind treatment phase: Participants received placebo once per month SC for 3 months during this phase.
  * Open-label treatment phase: After completion of double-blind phase, participants could enter open-label treatment phase where they received 240 mg loading dose of galcanezumab SC (2 injections of 120 mg) in the first month followed by 120 mg per month for 2 months.
  * Follow-up phase: After completion or discontinuation from double-blind or open-label treatment phases, participants entered follow-up phase where they were observed for 4 months. No treatments administered.
- Galcanezumab 120mg: * Double-blind treatment phase: Participants received 240 mg loading dose of galcanezumab SC (2 injections of 120 mg) in the first month followed by 120 mg per month for 2 months.
  * Open-label treatment phase: After completion of double-blind phase, participants could enter open-label treatment phase where they continued to receive 120 mg galcanezumab SC per month for 3 months.
  * Follow-up phase: After completion or discontinuation from double-blind or open-label treatment phases, participants entered follow-up phase where they were observed for 4 months. No treatments administered.
Period: Double-Blind Treatment Phase
Arm/Group | Placebo | Galcanezumab 120mg
Started | 259 | 261
Received at Least One Dose of Study Drug | 259 | 261
Completed | 242 | 245
Not Completed | 17 | 16
Not completed — Adverse Event | 0 | 6
Not completed — Protocol Violation | 1 | 1
Not completed — Pregnancy | 2 | 1
Not completed — Withdrawal by Subject | 13 | 5
Not completed — Physician Decision | 1 | 3
Period: Open-Label Treatment Phase
Arm/Group | Placebo | Galcanezumab 120mg
Started | 241 (Participants from double-blind treatment phase had the option to enter the open-label treatment phase or proceed directly to the follow-up phase.) | 243 (Participants from double-blind treatment phase had the option to enter the open-label treatment phase or proceed directly to the follow-up phase.)
Completed | 234 | 232
Not Completed | 7 | 11
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Pregnancy | 1 | 0
Period: Follow-up Phase
Arm/Group | Placebo | Galcanezumab 120mg
Started | 243 (Participants from double-blind or open-label treatment phases entered the follow-up phase.) | 247 (Participants from double-blind or open-label treatment phases entered the follow-up phase.)
Entered From Double-blind Treatment Phase | 7 | 11
Entered From Open-Label Treatment Phase | 236 | 236
Completed | 236 | 238
Not Completed | 7 | 9
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Protocol Violation | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Galcanezumab 120 mg | Total
Number analyzed (Participants) | 259 | 261 | 520
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.80 (9.83) | 37.20 (9.33) | 37.00 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 188 | 384
  Male | 63 | 73 | 136
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 239 | 239 | 478
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 22 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 198 | 198 | 396
  India | 41 | 41 | 82
  Russia | 20 | 22 | 42
Monthly Migraine Headache Days (MHD) [Mean (Standard Deviation); unit: days per month] | 8.34 (2.70) | 8.16 (2.83) | 8.25 (2.76)

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days (MHDs) During the Double-blind Treatment Phase.
Description: MHD is a calendar day on which a migraine or probable migraine (a headache missing 1 of the migraine features) occurred. Per International Headache Society [IHS] International Classification of Headache Disorders 3rd edition [ICHD-3], migraine is defined as a headache, with or without aura, of ≥30 minutes duration with the following required features (A) At least 2 of the following headache characteristics: Unilateral location; Pulsatile quality; Moderate or severe pain intensity; Aggravation by or causing avoidance of routine physical activity (B) During headache at least 1 of the following: Nausea and/or vomiting; Photophobia and phonophobia. Overall mean is derived from the average of months 1 to 3 with Least square (LS) mean change calculated using mixed model repeat measures (MMRM) model with fixed categorical effects of treatment, country, month, and treatment-by-month interaction, and the continuous fixed covariates of baseline value and baseline value-by-visit interaction.
Time Frame: Baseline, 3 Months
Population: All randomized participants who received at least one dose of study drug and had baseline, at least one non-missing post baseline value.
Measure: Least Squares Mean (Standard Error); unit: days per month
Groups:
- Placebo - Double-Blind Treatment Phase: Participants received placebo once per month SC for 3 months.
- Galcanezumab 120mg - Double-Blind Treatment Phase: Participants received 240 mg loading dose of galcanezumab SC (2 injections of 120 mg) in the first month followed by 120 mg per month for 2 months.
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 258 | 260
days per month | -1.99 (0.23) | -3.81 (0.23)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean Difference = -1.82, 95% CI 2-sided [-2.32 to -1.32], Standard Error of Mean 0.26

2. Secondary Outcome: Overall Mean Percentage of Participants With ≥30%, ≥50%, ≥75%, 100% Reduction From Baseline in Monthly Migraine Headache Days (MHDs) During the Double-blind Treatment Phase.
Description: Participant having:
  * 30% or greater reduction in the total number of MHDs relative to baseline in a 30-day period is considered to have 30% response rate to treatment or "30% responder."
  * 50% or greater reduction in the total number of MHDs relative to baseline in a 30-day period is considered to have 50% response rate to treatment or "50% responder."
  * 75% or greater reduction in the total number of MHDs relative to baseline in a 30-day period is considered to have 75% response rate to treatment or "75% responder."
  * 100% reduction in the total number of MHDs relative to baseline in a 30-day period is considered to have 100% response rate to treatment or "100% responder." Overall mean is derived from the average of months 1 to 3 using generalized linear mixed model (GLIMMIX) with the fixed categorical effects of treatment, month, and treatment-by-month interaction, as well as the continuous, fixed covariate of baseline value.
Time Frame: 3 Months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage of participants
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 258 | 260
Percentage of participants
  30% responder | 50.3 (2.4) | 73.0 (2.1)
  50% responder | 32.9 (2.3) | 54.9 (2.4)
  75% responder | 12.7 (1.6) | 29.2 (2.1)
  100% responder | 3.9 (0.9) | 11.9 (1.4)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; 30% responder; Test type: Superiority; p < .0001, GLIMMIX; Odds Ratio (OR) = 2.674, 95% CI 2-sided [2.010 to 3.557]
Statistical Analysis 2: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; 50% responder; Test type: Superiority; p < .0001, GLIMMIX; Odds Ratio (OR) = 2.481, 95% CI 2-sided [1.869 to 3.293]
Statistical Analysis 3: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; 75% responder; Test type: Superiority; p < .0001, GLIMMIX; Odds Ratio (OR) = 2.824, 95% CI 2-sided [2.007 to 3.972]
Statistical Analysis 4: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; 100% responder; Test type: Superiority; p < .0001, GLIMMIX; Odds Ratio (OR) = 3.309, 95% CI 2-sided [1.989 to 5.504]

3. Secondary Outcome: Overall Mean Change From Baseline in the Role Function-Restrictive Domain Score of the Migraine-Specific Quality-of-Life Questionnaire Version 2.1 (MSQ v2.1) During the Double-blind Treatment Phase.
Description: MSQ v2.1 is a self-administered instrument that was developed to address physical, emotional limitations of specific concern to individuals with migraine. It consists of 14 items that address 3 domains: Role Function-Restrictive (items 1-7), Role Function- Preventive (items 8-11) and Emotional Function (items 12-14). All item responses ranges from 1 (none of the time) to 6 (all of the time). Total raw scores for each domain is the sum of the raw scores of each item in that domain. After the total raw score is computed for each domain, they are transformed to a 0-100 scale with higher scores indicating a better health status & a positive change in scores reflecting functional improvement. Overall mean is derived from the average of months 1 to 3 with LS mean change calculated using MMRM model with fixed categorical effects of treatment, country, month, and treatment-by-month interaction, and the continuous fixed covariates of baseline value and baseline value-by-visit interaction.
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 248 | 260
score on a scale | 13.94 (0.88) | 21.01 (0.85)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean Difference = 7.07, 95% CI 2-sided [5.20 to 8.95], Standard Deviation 0.95

4. Secondary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days Requiring Medication for the Acute Treatment of Headache During the Double-blind Treatment Phase.
Description: Number of monthly migraine headache days requiring medication for the acute treatment of headache is defined as the number of calendar days in a 30-day period on which migraine or probable migraine occurs and acute medication is used. Overall mean is derived from the average of months 1 to 3 with LS mean change calculated using MMRM model with fixed categorical effects of treatment, country, month, and treatment-by-month interaction, and the continuous fixed covariates of baseline value and baseline value-by-visit interaction.
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days per month
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 258 | 260
days per month | -0.71 (0.22) | -2.49 (0.22)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean Difference = -1.78, 95% CI 2-sided [-2.25 to -1.31], Standard Error of Mean 0.24

5. Secondary Outcome: Overall Mean Change From Baseline in the Number of Monthly Headache Days During the Double-blind Treatment Phase.
Description: Number of monthly headache days is the number of calendar days in a 30-day period on which a headache occurs. Overall mean is derived from the average of months 1 to 3 with LS mean change calculated using MMRM model with fixed categorical effects of treatment, country, month, and treatment-by-month interaction, and the continuous fixed covariates of baseline value and baseline value-by-visit interaction.
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days per month
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 258 | 260
days per month | -2.09 (0.24) | -3.91 (0.24)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean Difference = -1.82, 95% CI 2-sided [-2.35 to -1.29], Standard Error of Mean 0.27

6. Secondary Outcome: Percentage of Participants Who Maintain 50% Response Criteria During the Double-blind Treatment Phase.
Description: Percentage of participants who maintained 50% response rate to treatment in all 3 months of the double-blind treatment phase.
Time Frame: Month 1 to Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 258 | 260
percentage of participants | 12.4 | 29.6
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 3.04, 95% CI 2-sided [1.92 to 4.81]

7. Secondary Outcome: Overall Mean Change From Baseline in Number of Monthly Migraine Attacks During the Double-blind Treatment Phase.
Description: Number of monthly migraine attacks is the number of sets of consecutive days with migraine or probable migraine separated by at least one migraine-free day in a 30-day period day. Overall mean is derived from the average of months 1 to 3 with LS mean change calculated using MMRM model with fixed categorical effects of treatment, country, month, and treatment-by-month interaction, and the continuous fixed covariates of baseline value and baseline value-by-visit interaction.
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: migraine attacks per month
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 258 | 260
migraine attacks per month | -1.57 (0.12) | -2.46 (0.12)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean Difference = -0.89, 95% CI 2-sided [-1.15 to -0.62], Standard Error of Mean 0.13

8. Secondary Outcome: Overall Mean Change From Baseline in Number of Monthly Migraine Headache Hours During the Double-blind Treatment Phase.
Description: Number of monthly migraine headache hours is the total number of headache hours in a 30-day period on days when a migraine or probable migraine occurs. Overall mean is derived from the average of months 1 to 3 with LS mean change calculated using MMRM model with fixed categorical effects of treatment, country, month, and treatment-by-month interaction, and the continuous fixed covariates of baseline value and baseline value-by-visit interaction.
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours per month
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 258 | 260
hours per month | -12.83 (1.98) | -31.72 (1.96)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean Difference = -18.88, 95% CI 2-sided [-23.21 to -14.56], Standard Error of Mean 2.20

9. Secondary Outcome: Overall Mean Change From Baseline in Number of Monthly Headache Hours During the Double-blind Treatment Phase.
Description: Number of monthly headache hours is the total number of headache hours in a 30-day period on which a headache occurred. Overall mean is derived from the average of months 1 to 3 with LS mean change calculated using MMRM model with fixed categorical effects of treatment, country, month, and treatment-by-month interaction, and the continuous fixed covariates of baseline value and baseline value-by-visit interaction.
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours per month
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 258 | 260
hours per month | -12.94 (2.06) | -32.18 (2.03)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean Difference = -19.24, 95% CI 2-sided [-23.73 to -14.75], Standard Error of Mean 2.29

10. Secondary Outcome: Overall Mean Change From Baseline in Severity of Migraine Headaches During the Double-blind Treatment Phase.
Description: Severity of Migraine Headache was measured on a headache severity scale ranging from 1 to 3 with 1=mild, 2=moderate, and 3=severe. The mean severity of migraine headache for each month will be calculated as: sum of severity of migraine headache days divided by number of migraine headache days. Overall mean is derived from the average of months 1 to 3 with LS mean change calculated using MMRM model with fixed categorical effects of treatment, country, month, and treatment-by-month interaction, and the continuous fixed covariates of baseline value and baseline value-by-visit interaction.
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 256 | 253
score on a scale | -0.03 (0.03) | -0.19 (0.03)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean Difference = -0.16, 95% CI 2-sided [-0.22 to -0.10], Standard Error of Mean 0.03

11. Secondary Outcome: Mean Change From Baseline in the Patient Global Impression of Severity (PGI-S) Score at Month 3 During the Double-blind Treatment Phase.
Description: PGI-S is a 7-point scale that measures participants own global impression of their illness severity. The participant was instructed as follows: "Considering migraine as a chronic condition, how would you rate your level of illness?" Response options range from 1 ("normal, not at all ill") to 7 ("extremely ill"). LS mean change was calculated using analysis of variance (ANCOVA) model with fixed categorical effects of treatment, country, and the continuous fixed covariates of baseline value and baseline value-by-visit interaction.
Time Frame: Baseline, Month 3
Population: All randomized participants who received at least one dose of study drug and had baseline value, non-missing post baseline value at month 3.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 238 | 252
score on a scale | -0.610 (0.0961) | -0.834 (0.0930)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p = 0.0284, ANCOVA; LS Mean Difference = -0.224, 95% CI 2-sided [-0.43 to -0.02], Standard Error of Mean 0.1021

12. Secondary Outcome: Mean Change From Baseline on the Migraine Disability Assessment Test (MIDAS) Total Score at Month 3 During the Double-blind Treatment Phase.
Description: The MIDAS was designed to quantify headache-related disability over a 3-month period. This instrument consists of 5 items that measures the impact that migraine headaches have on migraineurs' life, including days of work/school missed, days with productivity at work/school reduced to half or more, days with household work missed, days with productivity in household work reduced to half or more, and days missed family/social/leisure activities. Each item has a numeric response range from 0 to 90 days; if days are missed from work/school or household work they are not counted as days with reduced productivity at work/school or household work. The numeric responses are summed to produce a total score ranging from 0 to 270. A higher value is indicative of more disability. LS mean change was calculated using ANCOVA model with fixed categorical effects of treatment, country, and the continuous fixed covariates of baseline value and baseline value-by-visit interaction.
Time Frame: Baseline, Month 3
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 238 | 252
score on a scale | -10.181 (3.0597) | -22.610 (2.9582)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p = 0.0001, ANCOVA; LS Mean Difference = -12.429, 95% CI 2-sided [-18.81 to -6.05], Standard Error of Mean 3.2484

13. Secondary Outcome: Percentage of Participants With Treatment Emergent Anti-Drug Antibodies (TE-ADA) During the Double-blind Treatment Phase.
Description: A TE-ADA evaluable participant is considered to be TE-ADA positive if the participant has at least one post baseline titer that is a 4-fold or greater increase in titer from baseline measurement. If baseline result is ADA Not Present, then the participant is TE ADA positive if there is at least one post baseline result of ADA Present with titer >= 20.
Time Frame: Baseline to Month 3
Population: All randomized participants who received at least one dose of study drug and had baseline, at least one non-missing post baseline ADA value.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 248 | 259
percentage of participants | 1.2 | 9.3

14. Secondary Outcome: Pharmacokinetics (PK): Serum Concentration of Galcanezumab During the Double-blind Treatment Phase.
Description: PK: Serum concentration of galcanezumab
Time Frame: Month 3
Population: All randomized participants who received at least one dose of galcanezumab and had evaluable serum concentrations.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 260
Nanogram per milliliter (ng/mL) | 14696 (5675)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To 10 months)
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
  Per protocol, AE analysis was planned per treatment regimen received in each study phase
Groups:
- Placebo - Double-Blind Treatment Phase: Participants received placebo once per month SC for 3 months during this phase.
- Placebo/Galcanezumab 120mg - Open-Label Treatment Phase: After completion of Placebo double-blind phase, participants had an option to enter open-label treatment phase where they received 240 mg loading dose of galcanezumab SC (2 injections of 120 mg) in the first month followed by 120 mg per month for 2 months.
- Galcanezumab 120mg/Galcanezumab 120mg - Open-Label Treatment Phase: After completion of Galcanezumab 120mg double-blind phase, participants had an option to enter open-label treatment phase where they continued to receive 120 mg galcanezumab SC per month for 3 months.
- Placebo - Follow-up: Participants entered follow-up phase from Placebo double-blind treatment phase and were observed for 4 months. No treatments administered.
- Galcanezumab 120mg - Follow-up: Participants entered follow-up phase from Galcanezumab 120mg double-blind treatment phase and were observed for 4 months. No treatments administered.
- Placebo/Galcanezumab 120mg - Follow-up: Participants entered follow-up phase from Placebo/Galcanezumab 120 mg open-label treatment phase and were observed for 4 months. No treatments administered.
- Galcanezumab 120mg/Galcanezumab 120mg - Follow-up: Participants entered follow-up phase from Galcanezumab 120mg/Galcanezumab 120mg open-label treatment phase and were observed for 4 months. No treatments administered.
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase | Placebo/Galcanezumab 120mg - Open-Label Treatment Phase | Galcanezumab 120mg/Galcanezumab 120mg - Open-Label Treatment Phase | Placebo - Follow-up | Galcanezumab 120mg - Follow-up | Placebo/Galcanezumab 120mg - Follow-up | Galcanezumab 120mg/Galcanezumab 120mg - Follow-up
All-Cause Mortality (participants affected / at risk) | 0/259 | 0/261 | 0/241 | 0/243 | 0/7 | 0/11 | 0/236 | 0/236
Serious Adverse Events (participants affected / at risk) | 3/259 | 2/261 | 9/241 | 3/243 | 0/7 | 0/11 | 3/236 | 4/236
Other Adverse Events (participants affected / at risk) | 29/259 | 32/261 | 12/241 | 7/243 | 0/7 | 0/11 | 0/236 | 0/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Double-Blind Treatment Phase (N=259) | Galcanezumab 120mg - Double-Blind Treatment Phase (N=261) | Placebo/Galcanezumab 120mg - Open-Label Treatment Phase (N=241) | Galcanezumab 120mg/Galcanezumab 120mg - Open-Label Treatment Phase (N=243) | Placebo - Follow-up (N=7) | Galcanezumab 120mg - Follow-up (N=11) | Placebo/Galcanezumab 120mg - Follow-up (N=236) | Galcanezumab 120mg/Galcanezumab 120mg - Follow-up (N=236)
Thymic cyst (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic outlet syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1/196 (1) | 0/188 (0) | 0/180 (0) | 0/175 (0) | 0 (0) | 0/8 (0) | 0/177 (0) | 0/173 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/196 (0) | 0/188 (0) | 1/180 (1) | 0/175 (0) | 0 (0) | 0/8 (0) | 0/177 (0) | 0/173 (0)
Borderline personality disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0/196 (0) | 0/188 (0) | 0/180 (0) | 1/175 (1) | 0 (0) | 0/8 (0) | 0/177 (0) | 0/173 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Double-Blind Treatment Phase (N=259) | Galcanezumab 120mg - Double-Blind Treatment Phase (N=261) | Placebo/Galcanezumab 120mg - Open-Label Treatment Phase (N=241) | Galcanezumab 120mg/Galcanezumab 120mg - Open-Label Treatment Phase (N=243) | Placebo - Follow-up (N=7) | Galcanezumab 120mg - Follow-up (N=11) | Placebo/Galcanezumab 120mg - Follow-up (N=236) | Galcanezumab 120mg/Galcanezumab 120mg - Follow-up (N=236)
Injection site pain (General disorders) | 16 (37) | 19 (47) | 6 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 13 (14) | 14 (15) | 6 (7) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT03963232/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT03963232/SAP_001.pdf